CLINICAL TRIAL: NCT05563584
Title: Super-Rehab: Can we Achieve Coronary Artery Disease Regression? (a Feasibility Study)
Brief Title: Super-Rehab: Can we Achieve Coronary Artery Disease Regression?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Collaborators: University of Bath (Other); University of Oxford (Other); University of Bristol (Other); National Institute for Health Research, United Kingdom (Other Government); North Bristol NHS Trust (Other); RUHX (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RUH Bath NHS SR CAD
Record Dates: First submitted 2022-01-04; First posted 2022-10-03 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; Metabolic Syndrome
Keywords: Lifestyle risk reduction; Exercise; Inflammation; Behavior modifications; Nutrition therapy; Diet; Feasibility studies; Cardiovascular disease
MeSH Terms: conditions — Coronary Artery Disease; Metabolic Syndrome; Risk Reduction Behavior; Motor Activity; Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Patients randomized to Usual Care or Super Rehab plus Usual Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients will continue Usual Care, which will include aspirin, a statin and routine lifestyle advice
- Super Rehab plus Usual Care (Experimental): 12-month Super Rehab programme plus Usual Care
  Interventions: Behavioral: Super Rehab

INTERVENTIONS:
Behavioral: Super Rehab — A 12-month healthcare-delivered lifestyle intervention involving exercise and nutritional support
  Arms: Super Rehab plus Usual Care

SUMMARY:
The Super Rehab: Can we Achieve Coronary Artery Disease Regression? (a feasibility study) proposes to test the use of a novel lifestyle intervention (Super Rehab), in addition to standard care, for patients with both coronary artery disease and metabolic syndrome. This is a feasibility study that will test study processes, enable optimisation of the intervention and provide data for power calculations to enable design of pivotal trials of the clinical effectiveness of Super Rehab.

DETAILED DESCRIPTION:
In this research we will study the feasibility of a randomised controlled trial (RCT) of a novel lifestyle intervention (Super Rehab), in addition to usual care, for patients with established coronary artery disease (CAD) and metabolic syndrome. Increasing evidence has shown that CAD can not only be stabilised, but can in fact regress with treatments that include lifestyle interventions.

This feasibility study will involve patients undergoing a clinically indicated coronary CT angiography (CCTA) scan who are found to have confirmed CAD with plaque causing a narrowing in at least one coronary artery of ≥25% of the lumen on their CTCA; have evidence of coronary inflammation (defined by an abnormal fat attenuation index (FAI) of > -70.1HU or with FAI score [relative to age and sex matched patients] ≥ 75th percentile in the left anterior coronary or right coronary artery or with FAI score ≥ 90th percentile in the circumflex coronary); have Metabolic Syndrome, defined as any 3 of: high abdominal waist circumference (≥94cm males, ≥80cm females), hypertension (≥130/85mmHg or on treatment), raised fasting glucose (≥5.6mmol/L or on diabetic treatment), low HDL (≤1mmol/L males, <1.3mmol/L females), and high triglycerides (>1.7mmol/L).

Participants will be randomised to either Super Rehab and Usual Care or to continue Usual Care only. Super Rehab includes a combination of separate 1:1 supervised high-intensity exercise and dietary advice sessions, and the whole programme lasts 12 months. Participants in both arms will undergo imaging, fitness, clinical tests (including blood tests), and complete questionnaires on four occasions during the study, alongside short interim and detailed end-of-study interviews.

The study will primarily assess key feasibility outcomes to guide a potential subsequent RCT, e.g. recruitment and retention rates and test the acceptability of the intervention and study processes. In addition, the study will provide baseline data for power calculations to support study design for the planned future RCT into the clinical effectiveness of Super Rehab in this patient group.

ELIGIBILITY:
Inclusion Criteria:

1. CCTA demonstrating coronary artery disease with plaque causing a narrowing in at least one coronary artery of ≥ 25% stenosis and a evidence of coronary inflammation (defined by an abnormal fat attenuation index (FAI; defined as FAI > -70.1HU or with FAI score [relative to age and sex matched patients] ≥ 75th percentile in the left anterior coronary or right coronary artery or with FAI score ≥ 90th percentile in the circumflex coronary)
2. Have Metabolic Syndrome, defined as any 3 of: high abdominal waist circumference (≥94cm males, ≥80cm females), hypertension (≥130/85mmHg or on treatment), raised fasting glucose (≥5.6mmol/L or on diabetic treatment), low HDL (≤1mmol/L males, <1.3mmol/L females), and high triglycerides (>1.7mmol/L).

Exclusion Criteria:

1. Coronary artery disease requiring revascularisation
2. Unstable angina
3. New York Heart Association class III/IV heart failure or severe left ventricular impairment
4. Severe valve disease
5. Significant cardiomyopathy (as assessed by screening Cardiologist)
6. Severe hypertension (defined as blood pressure >180/120mmHg)
7. Uncontrolled cardiac arrhythmia
8. Previous aortic dissection
9. Recent acute pulmonary embolus deep vein thrombosis, stroke or transient ischaemic attack
10. Severe autonomic or peripheral neuropathy
11. Acute systemic illness or fever
12. Significant acute or chronic renal failure
13. Pulmonary fibrosis or interstitial lung disease
14. Physically unable to participate in exercise
15. Previous myocardial infarction or coronary re-vascularisation
16. Severe coronary calcification that precludes assessment of the coronary lumen on CCTA
17. A clinically significant ECG abnormality at the screening visit, which in the opinion of the screening Cardiologist exposes the subject to risk by enrolling in the trial
18. Pregnant or breastfeeding
19. Current participation in another intervention based research study
20. Inability to fully understand the verbal and written descriptions of the study and the instructions provided during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Establish recruitment rate | Week 0
  A key feasibility outcome for a potential future randomised controlled trial will be to establish recruitment rates: defined as the proportion of eligible patients who accept the invitation to participate in the study.
Establish retention rate | Month 15
  A key feasibility outcome for a potential future randomised controlled trial will be to examine retention: defined as the proportion of recruited participants who complete the study.
Establish adherence | Month 12
  A key feasibility outcome for a potential future randomised controlled trial will be to examine adherence: defined as, for participants in the intervention arm, the proportion of offered sessions completed.
Assess acceptability of the intervention | Month 12
  A key feasibility outcome for a potential future randomised controlled trial will be to examine the acceptability of the intervention (Super Rehab) to participants and clinicians. This will be assessed qualitatively by an end of study interview.
Assess acceptability of the study design | Month 15
  A key feasibility outcome for a potential future randomised controlled trial will be to examine the acceptability of the study design. This will be assessed qualitatively by an end of study interview.

SECONDARY OUTCOMES:
Evaluate data collection procedures | Month 15
  To confirm that all data collection procedures (clinical, intervention and health economic data points) are achievable. This will be assessed as a percentage of the total number data-points we attempt to collect.
Assess the use of routine clinical data (combination of body mass index and HbA1c) for identifying coronary artery disease patients with metabolic syndrome | Month 15
  The percentage of patients recruited who meet international consensus metabolic syndrome diagnostic criteria that have a body mass index >28kg/m2 and an HbA1c >42mmol/mol.
Establish preliminary data for coronary artery disease regression with this intervention assessed with the peri-coronary fat attenuation index | Month 12
  To obtain preliminary data for coronary artery disease regression with Super Rehab when assessed with peri-coronary fat attenuation index (mean change in control vs intervention arms), to inform power calculations for a future randomised controlled trial.
Establish key characteristics required in intervention delivery | Month 15
  A qualitative analysis of interviews with the study Patient Advisory Group will report the key characteristics required in the intervention (Super Rehab) delivery for a successful future study.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal United Hospitals Bath NHS Foundation Trust, Bath, United Kingdom

REFERENCES:
- See also: Research team website outlining research goals — http://www.ruh.nhs.uk/SuperRehab